CLINICAL TRIAL: NCT04184531
Title: An Observational, Clinical Study to Collect the Medical Data in Order to Determine the Craniofacial Characteristics Through Phenotypic Analysis on Children With Sensenbrenner Treated/Followed at the Hôpital Femme Mère Enfant From 2005
Brief Title: Sensenbrenner Clinical Study
Acronym: Sensenbrenner
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: Sensenbrenner_2019
Record Dates: First submitted 2019-11-22; First posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Sensenbrenner Syndrome
Keywords: Sensenbrenner Syndrome; phenotypic analysis; craniofacial characteristics
MeSH Terms: conditions — Cranioectodermal Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with Sensenbrenner Syndrome: Children with Sensenbrenner followed from 2005. Variable phenotype related to the mutation gene will be analysed to determine some possible prognostic factors of the risk of developing end-stage kidney disease.
  Interventions: Other: Medical Data Collect

INTERVENTIONS:
Other: Medical Data Collect — It is a retrospective clinical study and we will collect only the medical data registered in our hospital software

SUMMARY:
Sensenbrenner syndrome, also known as cranioectodermal dysplasia (CED), is a rare autosomal-recessive disorder belonging to the ciliopathy group of diseases. It is characterized by a facial dysmorphism, abnormal bone development and ectodermal defects including dental anomalies. CED is a heterogeneous condition with significant phenotypic and molecular variability, whose spectrum may include cases of renal impairment, hepatic fibrosis, retinitis pigmentosa and/or brain anomalies. In many cases, patients develop chronic kidney disease (CKD) due to nephronophthisis between 2 and 6 years of age. The aim of this retrospective study is to better understand the characteristics of this syndrome and to find prognostic factors of CKD. We make the hypothesis that an early diagnosis of the syndrome would lead to a better global management of patients (quality of life, delayed onset of end-stage renal disease).

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls.
* Aged 3 to 18 years old.
* Subjects with a Sensenbrenner's syndrome diagnosis and followed from 2005
* Parents/ legal guardian must provide non opposition prior to participation in the study

Exclusion Criteria:

* Patients whose parents / legal guardian have object to using the data usually collected for care

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with Sensenbrenner syndrome
Sampling Method: Non-Probability Sample
Enrollment: 4 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of renal impairment of 4 patients with Sensenbrenner identified with WDR19 and WDR35 mutations, through measurement of level of creatinine in the urine. | The result of Creatinine in children with Sensenbrenner syndrome will be collected though study completion an average of 1 year.
  In many cases, patients with this syndrome develop chronic kidney disease (CKD) due to nephronophthisis between 2 and 6 years of age. Nephronophthisis is characterized by decreased urine concentration ability, chronic tubulointerstitial nephritis, cystic kidney disease and progression towards end-stage kidney disease (ESKD). In this study, we would analyze the renal phenotypes through the level of Creatinine in the urine to detect early-stage kidney disease. All the data will be collected from the patient medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme-Mère-Enfant, Bron, France